CLINICAL TRIAL: NCT03827746
Title: The Effect of Kinesiophobia on Physical Activity, Balance and Falling in Parkinson's Disease Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Kültür University (Other)
Collaborators: Marmara University (Other); Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Ertürk, Research assistant, Istanbul Kültür University
Other Study IDs: 09.2017.226
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease; Kinesiophobia; Physical Activity; Balance; Falling
Keywords: Parkinson's Disease, Kinesiophobia, Physical Activity, Balance, Falling
MeSH Terms: conditions — Parkinson Disease; Kinesiophobia; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tampa Kinesiophobia Scale, Berg-Balance Test, International Physical Activity Questionnaire-Short Form, Falls Efficacy Scale — Tampa Kinesiophobia Scale: The TSK is a 17-item self report checklist using a 4-point Likert scale that was developed as a measure of fear of movement or (re)injury.
  Berg-Balance Test: 14-item scale designed to measure balance of the older adult in a clinical setting.
  International Physical Activity Questionnaire-Short Form: This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
  Falls Efficacy Scale: A 16- item self-administered questionnaire designed to assess fear of falling in mainly older population

SUMMARY:
The kinesiophobia; defined as irrational fear of movement, which may occur after painful injury and reduce physical activity. It develops the idea that movement in individuals will cause re-injury and cause additional pain to existing pain. Studies have shown that this situation leads to a decrease in physical fitness, avoidance of activity, decrease in quality of life and even depression in the long term. It is known that functional problems such as balance problems and decrease in physical activity level occur in patients with Parkinson's disease. However, in the literature, there is no study investigating the presence of kinesiophobia in patients with Parkinson's disease. Therefore, the aims of our study were to 1) determine the presence / absence of kinesiophobia in patients with Parkinson's disease 2) determine the relationship between kinesiophobia and falling, balance, physical activity level in the presence of kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Parkinson's disease according to the criteria of United Kingdom Brain Bank and diagnosed as Parkinson's disease by neurologist
* According to Hoehn-Yahr scale 1-3
* Mini-Mental Test score 24 and above

Exclusion Criteria:

* Another disease that will prevent walking
* Visual impairment and vestibular dysfunction
* Cognitive impairment

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consisted of patients with Parkinson's disease who were in 1-3 stages according to Hoehn-Yahr Scale.
  The sample consisted of 60 patients who applied to Istanbul University Cerrahpaşa Medical Faculty Neurology Department Movement Disorders Unit, complied with the inclusion criteria, read the information form and signed an informed consent form.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TSK) | 10 minutes
  It is a 17-item self report checklist using a 4-point Likert scale
Berg-Balance Test | 15-20 minutes
  14-item scale designed to measure balance of the older adult in a clinical setting. Scoring: A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56 41-56 = low fall risk 21-40 = medium fall risk 0 -20 = high fall risk
Falls Efficacy Scale | 5-7 minutes
  It is a 10 item scale where each item is rated on a scale of 1-10. A score of 10 signifies no confidence in these activities; a score of 1 indicates confidence. Out of a total score of 100, a score of 70 or above indicates the individual has a fear of falling.
International Physical Activity Questionnaire - Short form | 5-10 minutes
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. Walking = 3.3 METs Moderate Intensity = 4.0 METs Vigorous Intensity = 8.0 METs Total MET-minutes/week = Walk (METs*min*days) + Mod (METs*min*days) + Vig (METs*min*days)
  1. Low: • No activity is reported OR • Some activity is reported but not enough to meet Categories 2 or 3. 2. Moderate: • 3 or more days of vigorous activity of at least 20 minutes per day OR • 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day OR • 5 or more days of any combination of walking, moderate-intensity or vigorousintensity activities achieving a minimum of at least 600 MET-minutes/week. 3. High: • Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week OR • 7 or more days of any combination of walki

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)